CLINICAL TRIAL: NCT04757987
Title: An Observational Study of Shared Variation and Reciprocal Influences: Distress, Immune Function and Pain in HIV.
Brief Title: An Observational Study of Distress, Immune Function, and Pain in HIV.
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Brigham and Women's Hospital (Other); University of Adelaide (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Victoria Madden, Senior lecturer, University of Cape Town
Other Study IDs: 764/2019; K43TW011442 (NIH)
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; HIV; Distress, Emotional; Immune System and Related Disorders; Central Sensitisation
Keywords: Chronic pain; HIV; Innate Immune Response; Mental health; Hyperalgesia, secondary
MeSH Terms: conditions — Chronic Pain; Psychological Well-Being; Hyperalgesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pain-free: Report persistent pain at enrolment
- Persistent pain: Report no pain at enrolment
  Interventions: Other: Pain

INTERVENTIONS:
Other: Pain — As above
  Groups: Persistent pain

SUMMARY:
This case-control study focuses on pain in HIV, which is common despite antiretroviral therapy and compromises quality of life, mental health and daily functioning. Specifically, it will investigate the relationships between psychosocial distress, inflammation and pain in HIV.

DETAILED DESCRIPTION:
We plan to recruit 100 people and follow them for 6 months, taking repeated measures. Participants who report persistent pain at enrolment will be assessed at 0 (baseline), 2, 4, and 6 months. Participants who report no pain at enrolment will be assessed at 0 (baseline) and 6 months. All participants will also be invited to participate in weekly remote assessment of selected self-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive with viral suppression
* report either persistent pain or no pain at enrolment

Exclusion Criteria:

* pregnancy
* acute psychiatric condition requiring urgent care
* cognitive impairment preventing full participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic in South Africa.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist 25-item questionnaire | Baseline
  Psychosocial distress
Provoked inflammatory response | Baseline
  Multiplex assay
Brief Pain Inventory | Baseline
  Pain intensity

SECONDARY OUTCOMES:
Secondary hyperalgesia (surface area) | Baseline assessment only
  Induced in a subgroup
Brief Pain Inventory | Baseline
  Pain locations

CONTACTS AND LOCATIONS:
Overall Officials: Victoria J Madden, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Community Health Clinic [name withheld due to risk to participants], [City Withheld Due to Risk to Participants], Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
The final dataset will include demographic, health history, psychological, and physiological data. An important priority when considering sharing of these data is participant confidentiality, particularly considering the stigma and personal social risk associated with HIV+ status in South Africa. If the data can be adequately stripped of identifiers so as to eliminate risk to participants, then the final, de-identified data set will be made available to qualified users through a data sharing platform, and subject to a sharing agreement that includes (1) a commitment to using the data only for research purposes and not to identify any individual participant; and (2) a commitment to securing the data using appropriate computer technology.

REFERENCES:
- [Derived] Madden VJ, Mqadi L, Arendse G, Bedwell GJ, Msolo N, Lesosky M, Hutchinson MR, Peter JG, Schrepf A, Parker R, Edwards RR, Joska JA. Provoked cytokine response is not associated with distress or induced secondary hyperalgesia in people with suppressed HIV. Pain. 2025 Dec 1;166(12):e830-e843. doi: 10.1097/j.pain.0000000000003748. Epub 2025 Aug 7. PMID 40788259
- [Derived] Madden VJ, Msolo N, Mqadi L, Lesosky M, Bedwell GJ, Hutchinson MR, Peter JG, Parker R, Schrepf A, Edwards RR, Joska JA. Study protocol: an observational study of distress, immune function and persistent pain in HIV. BMJ Open. 2022 Jun 3;12(6):e059723. doi: 10.1136/bmjopen-2021-059723. PMID 36691234